CLINICAL TRIAL: NCT05706792
Title: Randomized Controlled Clinical Trial to Evaluate the Effectiveness of the Nordic Sensi Chair in the Treatment of Dementia Behavioral Disorders (NSC-DEMEN Study)
Brief Title: Effectiveness of the Nordic Sensi Chair in the Treatment of Dementia Behavioral Disorders (NSC-DEMEN)
Acronym: NSC-DEMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Principal Investigator, Jose-Maria Garcia-Alberca, MD, PhD, Director of the Instituto Andaluz de Neurociencia (IANEC), 17 Álamos Street, 29012 Málaga, Spain, Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NSC-DEMEN Study
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Dementia
Keywords: Dementia; Behavioral symptoms of dementia; Dementia care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This was a 16-week randomized, parallel, single-blind, controlled, clinical trial. After assessments for eligibility patients were randomly assigned to two groups of equal size: a treatment group that received three times a week one session per day of 20 minutes in the NSC Relax for relaxation program and a control group that did not participate in the activity mentioned for the treatment group, but received, at the same time and duration, the care and activities that were part of the daily routines of the center.
  The 16-week study extension included a first pre-treatment period of 2 weeks' duration prior to the start of the intervention to establish the baseline, followed by a second 12-week treatment period with the use of the NSC and, finally, a third post-treatment period conducted 2-week after completion of the intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic Sensi Chair (Experimental): Participants received three times a week one session per day of 20 minutes in the Relax for deep relaxation program of the Nordic Sensi Chair.
  Interventions: Device: Nordic Sensi Chair
- Standard of care (No Intervention): Participants did not participate in the Nordic Sensi Chair sessions, but received, at the same time and duration, the care and activities that were part of the daily routines of the center, including group sessions of cognitive stimulation, training in activities of daily living or communication training.

INTERVENTIONS:
Device: Nordic Sensi Chair — The Nordic Sensi Chair is an electrically operated rocking chair with built-in MusiCure music composed by Niels Eje. It is equipped with an integrated audio system with music recording based on more than 15 years of research on the calming and mentally stimulating effect of sound. The Nordic Sensi Chair has three different programs: Relax for deep relaxation, Refresh for recovery and Comfort for gentle relaxation. A 5 kg fiber blanket increases the feeling of security and relaxation, while helping users to perceive their own body. In addition to musical programming, the Nordic Sensi Chair provides predefined tactile stimulation and rocking motion, for a relaxing multi-sensory experience. All settings can be easily customized at the touch of a button. For the purposes of this study, the NSC deep relaxation program (Relax Program) was used.
  Arms: Nordic Sensi Chair

SUMMARY:
The main objective of this study is to evaluate the effectiveness of the Nordic Sensi® Chair (NSC) in the management of behavioral symptoms of dementia (BPSD) in real clinical practice in people with dementia admitted to nursing homes. The secondary objective of the present study is to assess its benefits on the performance of the daily work activities of care staff.

Although over time the BPSD have been treated predominantly with pharmacological measures, there is now sufficient scientific evidence to support the use of non-pharmacological therapies (NPT) for their management.Within this context, only a few studies have evaluated the use of rocking chairs for people with dementia. Modern rocking chairs may be suitable for long-term care because rocking, a rhythmically repeated movement, can contribute to psychosocial wellbeing .

In this regard, it is a focus of attention to consider the therapeutic role of the Nordic Sensi® Chair in the treatment of BPSD based on its ability to offer patients a sensory experience that brings the benefits of music therapy, therapeutic tactile stimulation, vestibular stimulation, and relaxation in an integrated way, especially those in nursing homes. The NSC is an electrically operated rocking chair with built-in MusiCure music. It is equipped with an integrated audio system with music recording. The NSC has three different programs: Relax for deep relaxation, Refresh for recovery and Comfort for gentle relaxation. In addition to musical programming, the NSC provides predefined tactile stimulation and rocking motion, for a relaxing multi-sensory experience.

In this study, the 20 minutes NSC deep relaxation program (Relax Program) will be used.

Participants are randomly assigned to two groups of equal size: a treatment group that receives three times a week one session per day of 20 minutes in the Relax for deep relaxation program of the NSC and a control group that does not participate in the activity mentioned for the treatment group, but receives, at the same time and duration, the care and activities that are part of the daily routines.

Although cognitive and functional symptoms have been the hallmarks of dementia, in recent years behavioral and psychological symptoms of dementia (BPSD) have become increasingly important. In all cases, BPSD is always one of the most important challenges that both the patient and their caregivers will face throughout the course of the disease.

DETAILED DESCRIPTION:
Objective The main objective of this study is to evaluate the effectiveness of the Nordic Sensi® Chair in the management of behavioral symptoms of dementia (BPSD) in real clinical practice in people with dementia (PwD) admitted to nursing homes. The secondary objective of the present study was to assess the benefits of the NSC on cognitive functioning and quality of life of patients as well as its benefits on the performance of the daily work activities of care staff.

Background Dementia is a neurodegenerative syndrome characterised by a progressive impairment of the cognitive and functional abilities that causes a huge social and human fracture. The number of people with dementia increases globally and according to population projections, if the current prevalence of dementia remains constant the number of people with dementia will rise to 82 million in 2030 and almost double in 2050.

In addition to the cognitive and functional deficits, behavioural and psychological symptoms of dementia (BPSD) are one of the most important challenges that both people with dementia (PwD) and their caregivers face throughout the course of the disease. BPSD consist of a heterogeneous group of symptoms such as depression, anxiety, delusions, hallucinations, irritability, disinhibition, agitation, aberrant motor behaviour, apathy or sleep and eating problems. BPSD results in decreased patient well-being, impaired quality of life, excess morbidity and hospital admission and cause a heavy burden on caregivers, often leading caregivers to make the decision to institutionalise. In nursing-homes BPSD can place a greater care staff stress and other residents.

BPSD management includes both pharmacological and nonpharmacological therapies. Medication is often used and many patients with late-stage dementia are treated with psychoactive drugs, although in many cases achieve only modest benefits in controlling symptoms while exposing patients to the risk of possible adverse events. On the contrary, nonpharmacological interventions are considered to have fewer undesirable effects making them safer options. Therefore, currently there is a consensus to consider nonpharmacological therapies as the first line treatment of BPSD with the exception of emergency situations or when symptoms have not responded effectively to non-pharmacological interventions.

There is a wide range of nonpharmacological approaches that have shown positive results for the management of BPSD from sensory to psychological and behavioural approaches including physical exercise, environmental interventions, music therapy, light therapy, aromatherapy, massage, multisensory stimulation, psycho-educational interventions for caregivers or care staff training. However, despite the public health problem posed by dementia, and more specifically the management of BPSD, there is a lack of well-designed studies evaluating the efficacy of the different nonpharmacological therapies.

Within this context, only a few studies have evaluated the use of rocking chairs for PwD. Modern rocking chairs may be suitable for long-term care because rocking, a rhythmically repeated movement, can contribute to psychosocial wellbeing. In this regard, it is a focus of attention to consider the therapeutic role of the Nordic Sensi® Chair (NSC) in the treatment of BPSD based on its ability to offer patients a sensory experience that brings the benefits of music therapy, therapeutic tactile stimulation, vestibular stimulation, and relaxation in an integrated way, especially those in nursing homes. This approach could facilitate the achievement of a balance between stimulation and sensory calm that would contribute to the effective management of BPSD.

The NSC (Wellness Nordic A/S, Humlebaek, Denmark) is an electrically operated rocking chair with built-in MusiCure music composed by Niels Eje. It is equipped with an integrated audio system with music recording based on more than 15 years of research on the calming and mentally stimulating effect of sound. The NSC has three different programs: Relax for deep relaxation, Refresh for recovery and Comfort for gentle relaxation. A 5 kg fiber blanket increases the feeling of security and relaxation, while helping users to perceive their own body. In addition to musical programming, the NSC provides predefined tactile stimulation and rocking motion, for a relaxing multi-sensory experience. All settings can be easily customized at the touch of a button.

The use of music in PwD, carried out on different stages of the disease, is based on the ancestral link between sounds and the human being and its potential to evoke emotions experienced throughout their lives, while generating states of calm and relaxation. This fact can be used to maximum benefit, as music can become a way of expressing their emotions in daily life, thus preventing the onset of anxious, agitated or even aggressive behaviour. Another way to increase the comfort of PwD is to provide tactile stimulation that could activate higher-order brain structures, such as the hypothalamus. As a result, patients would feel less anxious and calmer. Vestibular stimulation is very powerful as a tool to help regulate arousal levels to enable self-calming and focused attention.

Study participants in this study are men and women with a diagnosis of dementia according to the criteria of the 11th edition of the International Classification of Diseases of the World Health Organization and/or probable Alzheimer´s disease (AD) according to the criteria of the National Institute on Aging Alzheimer's Association workgroups (NIA/AA). Patients were recruited from two nursing homes specialized in dementia care: Centro Residencial Almudena (Rincón de la Victoria, Málaga, Spain) and Residencia DomusVi Fuentesol (Alhaurín de la Torre, Málaga, Spain). Patients included in the study are clinically defined in stages 4 to 7 of the Reisberg Global Deterioration Scale (GDS).

Considering the variability reported in the literature of the clinical assessment instruments used in the present study, it was anticipated that a sample of 70 subjects (35 in each of the two groups) would allow detection, with 80% power and an anticipated effect size of 0.5, for the primary efficacy variable NPI-NH of a statistically significant difference in the mean of 2.5 points or more between the two study groups, assuming a standard deviation of 1.5 points.

The study includes the evaluation of care staff from both nursing homes who participated in the direct provision of care to the participating PwD. The degree to which the presence of BPSD disturbed the normal development of their professional activities is assessed.

The study protocol was approved by the Málaga Research Ethics Committee (NSC-DEMEN study protocol approved on April 25, 2022). A written informed consent was signed by patients who were able to give or their legal representative. Informed consent was also requested from care staff who participated in the study. The study followed the ethical standards adopted by the Declaration of Helsinki in its latest version (Fortaleza, Brasil, 2013) and was conducted in accordance with the standards of Good Clinical Practice, as described in the Tripartite Harmonized Standards of the International Conference on Harmonisation for Good Clinical Practice 1996.

Study design This was a 16-week randomized, parallel, single-blind, controlled, clinical trial (RCT). After assessments for eligibility PwD were randomly assigned to two groups of equal size: a treatment group that received three times a week one session per day of 20 minutes in the Relax for deep relaxation program of the NSC and a control group that did not participate in the activity mentioned for the treatment group, but received, at the same time and duration, the care and activities that were part of the daily routines of the center, including group sessions of cognitive stimulation, training in activities of daily living or communication training. The research team evaluating the study results was blinded to the group assigned to the patients. An anonymized data base was generated. The safety of the intervention was closely monitored.

The 16-week study extension included a first pre-treatment period of 2 weeks' duration prior to the start of the intervention to establish the baseline, followed by a second 12-week treatment period with the use of the NSC and, finally, a third post-treatment period conducted 2-week after completion of the intervention. Participant assessments were conducted at four time points: at baseline, at weeks 6 and 12 of the treatment period, and at week 16 after the washout period.

Upon entry into the study, PwD who met the inclusion criteria were randomized to the treatment group or the control group. Randomization was carried out by blocks generating random numbers with repetition, one per block. Randomization numbers were assigned sequentially for all study participants.

Intervention For the purposes of this study, the NSC deep relaxation program (Relax Program) was used. The Relax Program lasts 20 minutes, during which the backrest descends to a semi-reclined position that is maintained throughout the program. The chair has also a footrest that can be raised and lowered. At the end of the program, the backrest returns to the sitting position. At the same time that the chair is rocking in a linear direction, the patient perceives the automatic relaxation music along with tactile stimulation on the back.

In both nursing homes, the treatment was carried out on weekdays, during the day shift. The chairs were placed in a quiet and separate space from the rest of the living areas intended exclusively for the treatment sessions, so there was no interference with the intervention. In each nursing home PwD were always introduced to the chair by the same nurse assistant who was specifically recruited and trained for the study. To facilitate the adaptation to the therapeutic process, participants were carefully introduced to the chair, e.g. just suggesting them sit down the first time, carefully rock the second time, start of the full program session the third time. During the treatment session, the nurse assistant remained seated next to the patient, ensuring that the user was relaxed and comfortable. Each PwD had their own schedule of rocking chair use throughout the study.

Outcomes measures Primary efficacy outcome was the Neuropsychiatric Inventory-Nursing Home (NPI-NH). Secondary efficacy outcomes were Cohen-Mansfield Agitation Inventory (CMAI) and Cornell Scale for Depression in Dementia (CSDD).

Statistical analysis A Mixed Effects Model Analysis for Repeated Measurements (MMRM) was carried out in order to evaluate changes in neuropsychiatric, cognitive, and functional scores and to handle missing value in some of the follow-up assessments. The effect of time (between the mean baseline measurements and each time point), treatment and treatment by time interactions were evaluated. All analyses were controlled for demographic and clinical characteristics that approached significance on univariate analysis. Post hoc analyses for multiple comparisons were conducted using Bonferroni´s correction. Cohen's d standardized effect sizes were calculated and defined as small d=0.20, medium d=0.50 and large d=0.80 [30].

The main efficacy analysis was based on the Intent-to-Treat (ITT) population using a Last Observation Carried Forward (LOCF) imputation. This ITT-LOCF population was pre-defined as all randomized patients who received at least one week of the Nordic Sensi® Chair treatment and had a baseline and at least one post-baseline assessment for the primary efficacy variable on treatment.

Statistical analysis was performed with a significance of p≤0.05. SPSS Statistics version 25.0 (IBM Corporation, Armonk, New York, USA) was used for the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a diagnosis of dementia according to the criteria of the eleventh edition of the International Classification of Diseases of the World Health Organization (ICD-11).
* The patients will be clinically defined in stages 5 to 7 of the Reisberg Global Deterioration Scale (GDS).
* All selected patients should have data on physical examination, neurological and psychiatric examination, as well as neuropsychological evaluation in their clinical history.
* Written informed consent signed by the patient or his/her legal representative

Exclusion Criteria:

* Presence of focal neurological signs.
* Presence of focal vascular signs such as infarcts, microhemorrhages, hematomas, strokes, normal pressure hydrocephalus.
* Significant neurological history, such as brain trauma, brain tumors....
* Patients with epilepsy or inflammatory brain disease.
* Severe systemic diseases such as hypothyroidism or chronic renal failure.
* Substance abuse.
* Absence of a reliable informant.
* Absence of a complete medical history to assess study variables.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Change in behavioral and psychological symptoms of dementia measured by the Neuropsychiatric Inventory Nursing Home. | Baseline, 6 week, 12 week, 14 week.
  The Neuropsychiatric Inventory Nursing Home is an instrument to be used by the nursing staff to evaluate neuropsychiatric symptoms in people with dementia in the nursing home setting. The NPI-NH is composed of 12 domains that rate the most frequent behavioral and psychological symptoms of dementia. If a symptom was present during the previous month, frequency (ranging from 1 to 4), severity (ranging from 1 to 3) and composite scores (frequency x severity, ranging from 1 to 144) were obtained. Higher scores mean greater severity of behavioural symptoms.

SECONDARY OUTCOMES:
Change in agitation measured by the Cohen-Mansfield Agitation Inventory. | Baseline, 6 week, 12 week, 14 week.
  The Cohen-Mansfield Agitation Inventory composed of 30 items that form four subscales: psychically aggressive behaviors, non-psychically aggressive behaviors, verbally aggressive behaviors and non-verbally aggressive behaviours. Higher scores mean greater severity of agitation.
Change in depression measured by the Cornell Scale for Depression in Dementia. | Baseline, 6 week, 12 week, 14 week.
  The Cornell Scale for Depression in Dementia is a 19-item semi structured interview designed to assess depression in people with dementia with scores above 10 indicating a possible depression and scores above 18 suggesting a definitive depression. Higher scores mean greater severity of depression.

OTHER OUTCOMES:
Change in cognitive function measured by the Severe Mini Mental State Examination. | Baseline, 14 week.
  The Severe Mini Mental State Examination assesses the cognitive deterioration in patients with and advanced dementia. It is composed of 10 items and the score can reach 30 points. Lower scores mean greater cognitive impairment.
Change in functional status measured by the Bedford Alzheimer Nursing-Severity Scale. scores at 14 weeks. | Baseline, 14 week.
  The Bedford Alzheimer Nursing-Severity Scale consists of 7 items with 4 categories that enables to discriminate changes in advanced phases of dementia. The score ranges from 7 (no impairment) to 28 (total impairment). It assesses the patient's ability to perform three daily activities (dressing, eating and mobility), their ability to speak, their ability to maintain visual contact, the regularity of their sleep-wake cycle and the state of their muscles. Higher scores mean greater functional impairment.
Change in quality of life measured by the Quality of Life in Late-stage Dementia. | Baseline, 14 week.
  The Quality of Life in Late-stage Dementia of 11 items and evaluates three domains: affective state, confort and basic activities of life. Score ranges from 11 to 55, with lower scores being the highest quality of life.
Change in care staff´s stress measured by the Occupational Disruptiveness subscale of the Neuropsychiatric Inventory-Nursing Home. | Baseline, 6 week, 12 week, 14 week.
  The Occupational Disruptiveness subscale of the Neuropsychiatric Inventory-Nursing Home assesses the grade of self-reported professional caregiver burden, occupational carer's burden. Caregivers rate to what extent this behaviour disrupts them and/or generate more work. Score ranges from 0 to 5 points for each of the behaviour evaluated. Higher scores mean greater occupational disruptiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Garcia-Alberca, MD, PhD, Principal Investigator — Instituto Andaluz de Neurociencia (IANEC), 17 Álamos Street, 29012 Málaga, Spain
Locations (1):
- Instituto Andaluz de Neurociencia, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD and datasets used and/or analyzed during the present study will be made available through the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and datasets used and/or analyzed during this study will be available 6 months after the publication of the results for 5 years
Access Criteria: At the present time, we do not have a public repository URL with a direct link to our data because we are still working on them. However, data supporting the findings of this study are available from the principal investigator. Data may be shared with researchers and institutions related to the research topic. We may share the study protocol, the informed consent form, and the data. The latter, will be available once we have analyzed the database. The access mechanism, for the moment, is through the principal investigator upon reasonable request.

REFERENCES:
- [Background] van der Linde RM, Dening T, Stephan BC, Prina AM, Evans E, Brayne C. Longitudinal course of behavioural and psychological symptoms of dementia: systematic review. Br J Psychiatry. 2016 Nov;209(5):366-377. doi: 10.1192/bjp.bp.114.148403. Epub 2016 Aug 4. PMID 27491532
- [Background] Rocca P, Leotta D, Liffredo C, Mingrone C, Sigaudo M, Capellero B, Rocca G, Simoncini M, Pirfo E, Bogetto F. Neuropsychiatric symptoms underlying caregiver stress and insight in Alzheimer's disease. Dement Geriatr Cogn Disord. 2010;30(1):57-63. doi: 10.1159/000315513. Epub 2010 Aug 5. PMID 20689284
- [Background] Wetzels RB, Zuidema SU, de Jonghe JF, Verhey FR, Koopmans RT. Determinants of quality of life in nursing home residents with dementia. Dement Geriatr Cogn Disord. 2010;29(3):189-97. doi: 10.1159/000280437. Epub 2010 Mar 6. PMID 20215750
- [Background] Bessey LJ, Walaszek A. Management of Behavioral and Psychological Symptoms of Dementia. Curr Psychiatry Rep. 2019 Jul 1;21(8):66. doi: 10.1007/s11920-019-1049-5. PMID 31264056
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Seitz DP, Brisbin S, Herrmann N, Rapoport MJ, Wilson K, Gill SS, Rines J, Le Clair K, Conn D. Efficacy and feasibility of nonpharmacological interventions for neuropsychiatric symptoms of dementia in long term care: a systematic review. J Am Med Dir Assoc. 2012 Jul;13(6):503-506.e2. doi: 10.1016/j.jamda.2011.12.059. Epub 2012 Feb 17. PMID 22342481
- [Background] Snyder M, Tseng Y, Brandt C, Croghan C, Hanson S, Constantine R, Kirby L. A glider swing intervention for people with dementia. Geriatr Nurs. 2001 Mar-Apr;22(2):86-90. doi: 10.1067/mgn.2001.115197. PMID 11326215
- [Background] Zhang Y, Cai J, An L, Hui F, Ren T, Ma H, Zhao Q. Does music therapy enhance behavioral and cognitive function in elderly dementia patients? A systematic review and meta-analysis. Ageing Res Rev. 2017 May;35:1-11. doi: 10.1016/j.arr.2016.12.003. Epub 2016 Dec 23. PMID 28025173
- [Background] Wood S, Cummings JL, Hsu MA, Barclay T, Wheatley MV, Yarema KT, Schnelle JF. The use of the neuropsychiatric inventory in nursing home residents. Characterization and measurement. Am J Geriatr Psychiatry. 2000 Winter;8(1):75-83. doi: 10.1097/00019442-200002000-00010. PMID 10648298
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Koder D, Hunt GE, Davison T. Staff's views on managing symptoms of dementia in nursing home residents. Nurs Older People. 2014 Nov;26(10):31-6. doi: 10.7748/nop.26.10.31.e638. PMID 25430844
- [Background] Gruber-Baldini AL, Boustani M, Sloane PD, Zimmerman S. Behavioral symptoms in residential care/assisted living facilities: prevalence, risk factors, and medication management. J Am Geriatr Soc. 2004 Oct;52(10):1610-7. doi: 10.1111/j.1532-5415.2004.52451.x. PMID 15450035
- [Background] Zucchella C, Sinforiani E, Tamburin S, Federico A, Mantovani E, Bernini S, Casale R, Bartolo M. The Multidisciplinary Approach to Alzheimer's Disease and Dementia. A Narrative Review of Non-Pharmacological Treatment. Front Neurol. 2018 Dec 13;9:1058. doi: 10.3389/fneur.2018.01058. eCollection 2018. PMID 30619031
- [Background] Krutter S, Schaffler-Schaden D, Essl-Maurer R, Wurm L, Seymer A, Kriechmayr C, Mann E, Osterbrink J, Flamm M. Comparing perspectives of family caregivers and healthcare professionals regarding caregiver burden in dementia care: results of a mixed methods study in a rural setting. Age Ageing. 2020 Feb 27;49(2):199-207. doi: 10.1093/ageing/afz165. PMID 31875879
- [Background] Sprangers S, Dijkstra K, Romijn-Luijten A. Communication skills training in a nursing home: effects of a brief intervention on residents and nursing aides. Clin Interv Aging. 2015 Jan 20;10:311-9. doi: 10.2147/CIA.S73053. eCollection 2015. PMID 25653513
- [Background] Burks HB, des Bordes JKA, Chadha R, Holmes HM, Rianon NJ. Quality of Life Assessment in Older Adults with Dementia: A Systematic Review. Dement Geriatr Cogn Disord. 2021;50(2):103-110. doi: 10.1159/000515317. Epub 2021 Jun 24. PMID 34167127
- [Background] Kim SK, Park M. Effectiveness of person-centered care on people with dementia: a systematic review and meta-analysis. Clin Interv Aging. 2017 Feb 17;12:381-397. doi: 10.2147/CIA.S117637. eCollection 2017. PMID 28255234
- [Background] Lee KH, Lee JY, Kim B. Person-Centered Care in Persons Living With Dementia: A Systematic Review and Meta-analysis. Gerontologist. 2022 Apr 20;62(4):e253-e264. doi: 10.1093/geront/gnaa207. PMID 33326573
- [Background] Harrell LE, Marson D, Chatterjee A, Parrish JA. The Severe Mini-Mental State Examination: a new neuropsychologic instrument for the bedside assessment of severely impaired patients with Alzheimer disease. Alzheimer Dis Assoc Disord. 2000 Jul-Sep;14(3):168-75. doi: 10.1097/00002093-200007000-00008. PMID 10994658
- [Background] Volicer L, Hurley AC, Lathi DC, Kowall NW. Measurement of severity in advanced Alzheimer's disease. J Gerontol. 1994 Sep;49(5):M223-6. doi: 10.1093/geronj/49.5.m223. PMID 8056941
- [Background] Weiner MF, Martin-Cook K, Svetlik DA, Saine K, Foster B, Fontaine CS. The quality of life in late-stage dementia (QUALID) scale. J Am Med Dir Assoc. 2000 May-Jun;1(3):114-6. PMID 12818023
- [Derived] Garcia-Alberca JM, de la Rosa MD, Solo de Zaldivar P, Ledesma M, Oltra E, Gris E, Ocejo O, Torrecilla J, Zafra C, Sanchez-Fernandez A, Mancilla T, Lopez-Romero M, Jerez R, Santana N, Lara JP, Barbancho MA, Blanco-Reina E. Effect of Nordic Sensi(R) Chair on Behavioral and Psychological Symptoms of Dementia in Nursing Homes Residents: A Randomized Controlled Trial. J Alzheimers Dis. 2023;96(4):1609-1622. doi: 10.3233/JAD-230391. PMID 38007648